CLINICAL TRIAL: NCT02332460
Title: Incidence, Risk Factors and Immunologic Mechanisms of Infusion Related Reactions in Patients With Chronic Inflammatory Disease Receiving Infliximab
Brief Title: Infusion Related Reactions in Patients Receiving Infliximab
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/1368
Record Dates: First submitted 2014-11-28; First posted 2015-01-06 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Chronic Inflammatory Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — immunological and biochemical biomarkers, autoimmune antibodies, antibodies to infliximab, allergy analysis, concentrations of drugs (Infliximab, Metothrexat, and Imurel), HLA type
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infliximab: Patients treated with Infliximab

SUMMARY:
Infliximab is the active ingredient in a drug currently sold by the trade names Remicade, Remsima and Inflectra. Infliximab neutralizes tumor necrosis factor (TNF) α, a chemical messenger (cytokine) in the immune system, and belongs to a class of drugs called "TNF inhibitors". 8-55% of patients receiving infliximab have an infusion reaction. Infusion reactions are unintended reactions that occur during infusion of the drug and up to 14 days after. The incidence varies widely in different studies and seems difficult to determine due to variations in reporting of reactions, different definitions of reactions and retrospective data collection. The aim of this study is to estimate the incidence of infusion related reactions and investigate risk factors and immunological mechanisms of infusion reactions to infliximab in patients with a chronic inflammatory disease.

DETAILED DESCRIPTION:
Background: Infliximab is the active ingredient in a drug currently sold by the trade names Remicade, Remsima and Inflectra. Infliximab neutralizes tumor necrosis factor (TNF) α, a chemical messenger (cytokine) in the immune system, and belongs to a class of drugs called "TNF inhibitors". This class of drug comprises effective, biological agents used in the treatment of chronic inflammatory diseases. The use of TNF inhibitors is increasing, and infliximab is the third bestselling drug by value in Norway in 2013. By being a recombinant monoclonal antibody with a murine region, infliximab is associated with infusion reactions. 8-55% of patients receiving infliximab have an infusion reaction. Infusion reactions are unintended reactions that occur during infusion of the drug and up to 14 days after. The incidence varies widely in different studies and seems difficult to determine due to variations in reporting of reactions, different definitions of reactions and retrospective data collection. Protective factors, risk factors and the causes of the reactions are not well known. Different treatment strategies are being used, but evidence of efficacy varies.

Aim: The aim of this study is to estimate the incidence of infusion related reactions and investigate risk factors and immunological mechanisms of infusion reactions to infliximab in patients with a chronic inflammatory disease.

Primary objective:

Estimate the incidence of infusion reactions in patients with chronic inflammatory disease receiving infliximab

Secondary objectives:

* Evaluate the correlation between infusion reactions and the formation of antibodies to infliximab.
* Identify individual risk factors for infusion reactions to infliximab.
* Identify immunological mechanisms of infusion reactions to infliximab.
* Identify immunomodulatory effects and immunological changes in the patients during treatment with infliximab.

Study population: The study will be a prospective, longitudinal study where all departments with patients starting infliximab or switching infliximab from one supplier to another in the Western Norway Health Region (Helse Vest RHF) are invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with Infliximab due to chronic inflammatory disease included before start of treatment
* Weight at least 15 kg
* Control groups which may be included for investigations of secondary outcomes: age, gender, disease matched patients not receiving infliximab, healthy blood donors, other patients receiving pneumococci and influenza vaccines

Exclusion Criteria:

* Patients not completing treatment within Health Region
* Patients not able to complete sampling procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be a prospective, longitudinal study where all departments with patients starting infliximab or switching infliximab from one supplier to another in the Western Norway Regional Health Authority (Helse Vest RHF) are invited to participate.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2015-02; Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
incidence of infusion reactions | participants will be followed for the duration of treatment, an expected average of 62 weeks

SECONDARY OUTCOMES:
antibodies to infliximab | followed for the duration of treatment, an expected average of 62 weeks
  Specific IgG and IgE against ifliximab
immunological mechanisms of infusion reactions to infliximab | baseline (before infusion), during reaction, 12-24 hours after reaction
  allergy tests, cytokines, complement
autoantibodies and other immunological changes in the patients during treatment with infliximab | followed for the duration of treatment, an expected average of 62 weeks
individual risk factors for infusion reactions to infliximab | baseline
  HLA type, allergic predisposition
antibodies to pneumococci and influenza | baseline and 6-8 weeks after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Torunn Apelseth, MD, PhD, Study Director — Laboratory of Clinical Biochemistry, Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No